CLINICAL TRIAL: NCT04737772
Title: A Brief Behavioral Intervention for Co-users of Marijuana (MJ) and Tobacco Among Smokers Calling State Quitlines
Brief Title: Project CheckUP: A Brief Behavioral Intervention for Quitline Callers Who Use Marijuana (MJ) and Tobacco
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consumer Wellness Solutions (Industry)
Collaborators: University of Washington (Other); SRI International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R34DA051051 (NIH)
Record Dates: First submitted 2021-01-12; First posted 2021-02-04 (Actual); Results first posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Smoking Cessation; Marijuana Use
Keywords: smoking cessation; marijuana use
MeSH Terms: conditions — Smoking Cessation; Marijuana Use

STUDY DESIGN:
Intervention Model Description: A single arm pilot followed by a 2 arm randomized control trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Quitline Treatment As Usual (TAU) (Active Comparator): State quitline treatment as usual
  Interventions: Behavioral: Behavioral: Quitline treatment as usual
- QL Marijuana Check-Up intervention (QL-MJCU). (Experimental): Newly developed intervention for co-users of marijuana and tobacco.
  Interventions: Behavioral: QL Marijuana Check-Up intervention (QL-MJCU)

INTERVENTIONS:
Behavioral: Behavioral: Quitline treatment as usual — TAU is state quitline treatment that may include coaching sessions, text messaging and access to the web-based program plus cessation medications and unlimited calls to the QL for support between sessions.
  Arms: Standard Quitline Treatment As Usual (TAU)
Behavioral: QL Marijuana Check-Up intervention (QL-MJCU) — QL Marijuana Check-Up intervention (QL-MJCU) was developed for non-treatment seeking MJ users and is based on Motivational Enhancement Therapy. Includes TAU (see standard quitline arm) with a trained coach plus a MJ assessment and Personalized Feedback Report (PFR).
  Arms: QL Marijuana Check-Up intervention (QL-MJCU).

SUMMARY:
Smoking cigarettes remains the number one preventable cause of death and disease in the US. Smokers who call tobacco quitlines and use marijuana struggle to quit tobacco due to the interactive effects of nicotine and marijuana. A recent study found that 25% of callers to state quitlines said they were using marijuana and 44% of those were interested in quitting or cutting back their marijuana use (in addition to wanting to quit smoking). The investigators propose to develop an integrated intervention for co-users of marijuana and tobacco to be delivered via state-funded quitlines. The investigators will incorporate key elements of an evidence-based brief behavioral intervention called 'The Marijuana Check-Up' into the tobacco quitline treatment. The investigators will evaluate the feasibility, acceptability and preliminary effects of the new intervention in a small randomized pilot study with 100 co-users recruited from four participating state quitlines. Outcomes measured at 3 months post randomization will include tobacco abstinence (biochemically verified) and days used marijuana. The investigators hypothesize that the intervention will: (1) be feasible to deliver (measured by coach treatment fidelity scores); (2) be acceptable to co-users (measured by enrollments into the study and call completion numbers); (3) increase tobacco cessation rates compared with standard quitline treatment; (4) increase co-users motivation to change MJ use; and (5) produce greater reduction in days using MJ compared with standard quitline treatment. The proposed brief behavioral intervention addressing co-use may increase quitline callers' chances of achieving and maintaining tobacco abstinence and increase participants' motivation to reduce marijuana use. As non-medicinal marijuana use becomes common and legal in more states, a low touch phone and web-based intervention for co-users of marijuana and tobacco could improve health outcomes for many. Findings will inform development of scalable public health intervention strategies for co-users easily implemented across quitlines.

DETAILED DESCRIPTION:
We proposed to adapt a brief motivational intervention for cannabis (CB)) users who call tobacco quitlines for help quitting tobacco. We plan to recruit 100 adult co-users of tobacco and CB from four state quitlines that have legalized non-medicinal CB user. Quitline registration staff screen participants for current use of CB and interest in learning about CB use. Interested co-users will then talk to a specially trained quit coach who will ask additional eligibility questions, obtain informed consent from eligible participants, conduct a baseline assessment, randomize individuals to one of two groups and deliver the first counseling session according to the assigned intervention. Randomization is automated using the pre-programmed random number table (stratified by state and gender) built into the Quitline coaching application. Individuals are randomly assigned to receive the standard Quitline or the integrated CB and quitline intervention. All participants receive the standard quitline treatment: 4-5 counseling sessions delivered over the phone, mailed materials, access to the text messaging and web-based program plus cessation medications (nicotine replacement therapy; NRT) and unlimited calls into the quitline for help between calls. Quit coaches will deliver the CB intervention during the tobacco quitline calls for the intervention group. Study participants complete surveys at baseline and 3-months. We will compare groups on treatment engagement (calls completed) and outcomes at 3 months (tobacco abstinence and change in days used CB). Our proposed sample size of 100 (50 per group) is sufficient to achieve our study aims of assessing the feasibility, acceptability and preliminary effectiveness of the new integrated intervention compared with standard quitline treatment.

ELIGIBILITY:
Inclusion Criteria:

* daily use of 5 or more tobacco cigarettes
* aged 21 and older
* recruited from participating state quitlines (AK, DC, OR, WA)
* provides an email address
* wants to quit tobacco in the next 30 days
* used cannabis on 9 or more days in the past 30 days

Exclusion Criteria

* unable to speak and read English
* have limited access to a telephone
* pregnant or post-partum (because they are not offered the standard QL program)
* self-reported schizophrenia
* all cannabis use is recommended by a doctor or other healthcare professional

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly M Carpenter, PhD, Principal Investigator — Consumer Wellness Solutions (Optum)
Locations (1):
- Optum, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carpenter KM, Walker DD, Mullis K, Berlin HM, Short E, Javitz HS, Carlini BH. Testing a Brief Quitline Intervention for Tobacco Cannabis Co-Users: A Randomized Controlled Pilot Study. Tob Use Insights. 2024 Jun 12;17:1179173X241261302. doi: 10.1177/1179173X241261302. eCollection 2024. PMID 38873657

RESULTS

PARTICIPANT FLOW:
Period: Phase 2 Study
Arm/Group | Standard Quitline Treatment As Usual (TAU) | QL Marijuana Check-Up Intervention (QL-MJCU).
Started | 53 | 54
Completed | 34 | 38
Not Completed | 19 | 16
Not completed — Lost to Follow-up | 15 | 15
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Did not take any coaching calls | 4 | 0
Period: Pilot Phase 1 of Study
Arm/Group | Standard Quitline Treatment As Usual (TAU) | QL Marijuana Check-Up Intervention (QL-MJCU).
Started | 0 | 12
Completed | 0 | 10
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Randomized but ineligible | 0 | 1

BASELINE CHARACTERISTICS:
Population: We had 1 participant in the experimental group who withdrew from the study and 4 participants in the control group who did not take any coaching calls; therefore, we did not analyze their data or include them in the final dataset.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Quitline Treatment As Usual (TAU) | QL Marijuana Check-Up Intervention (QL-MJCU). | Total
Number analyzed (Participants) | 49 | 53 | 102
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.4 (14.3) | 52.9 (13.0) | 51.7 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 51
  Male | 24 | 27 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 49 | 51 | 100
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 7 | 9 | 16
  White | 37 | 38 | 75
  More than one race | 3 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 49 | 53 | 102
Poitive Screening for Depression (PHQ-2) [Count of Participants; unit: Participants] | 20 | 14 | 34
POsitive Screening for Anxiety (GAD-2) [Count of Participants; unit: Participants] | 20 | 14 | 34
PSS-4 [Mean (Standard Deviation); unit: units on a scale] — Participants are asked 4 questions regarding perceived stress (PSS-4=Perceived Stress Scale 4) on a scale from 0-4 with a total score of "0" being the lowest (best outcome) and a total score of "16" being the highest (worse outcome).
  units on a scale | 6.8 (3.5) | 5.7 (2.7) | 6.2 (3.2)
Cigarettes Per Day [Mean (Standard Deviation); unit: number of cigarettes per day] | 17.4 (8.1) | 15.2 (7.2) | 16.3 (7.7)
Time to First Cigarette Use [Count of Participants; unit: Participants] — Many research studies have reported that the time to first cigarette (TTFC) of the day is one of the strongest indicators of nicotine dependence.
  Participants
    Within 5 Minutes | 14 | 20 | 34
    6-30 minutes | 26 | 22 | 48
    31-60 Minutes | 7 | 6 | 13
    More than 60 Minutes | 2 | 5 | 7
Days of Cannabis Use Within Last 30 Days [Mean (Standard Deviation); unit: Days] | 25.7 (6.8) | 24.0 (7.4) | 24.8 (7.1)
Daily Cannabis Use (20+ Days in Last 30 Days) [Count of Participants; unit: Participants] | 41 | 39 | 80
Cannabis Use Disorder Identification Test [Mean (Standard Deviation); unit: units on a scale] — The CUDIT (Cannabis Use Disorder Identification Test) was designed for self-administration and is scored by adding each of the 8 items. Questions 1-7 are scored on a 0-4 scale. Question 8 is scored 0, 2 or 4. Scores of 8 or more indicate hazardous cannabis use, while scores of 12 or more indicate a possible cannabis use disorder for which further intervention may be required.
  units on a scale | 10.2 (4.9) | 10.1 (4.4) | 10.1 (4.7)
Readiness to Quit Cannabis [Mean (Standard Deviation); unit: units on a scale] — The Readiness to Quit Cannabis measures an individual's perceived readiness to quit cannabis use based on a scale from 1-10 with 1 being not ready at all and 10 being very ready.
  units on a scale | 3.4 (3.2) | 3.3 (3.2) | 3.3 (3.2)
Readiness to Reduce Cannabis [Mean (Standard Deviation); unit: units on a scale] — The Readiness to Reduce Cannabis measures an individual's perceived readiness to reduce cannabis use based on a scale from 1-10 with 1 being not ready at all and 10 being very ready.
  units on a scale | 4.2 (3.3) | 4.1 (3.3) | 4.2 (3.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Calls Completed
Description: Number of calls completed (collected during treatment and finalized at end of study)
Time Frame: from program enrollment up to 3 months post-enrollment
Population: 4 TAU participants did not receive coaching calls and 1 QL-MJCU participant withdrew from the study; therefore their outcomes data were not analyzed
Measure: Number; unit: Total number of calls
Arm/Group | Standard Quitline Treatment As Usual (TAU) | QL Marijuana Check-Up Intervention (QL-MJCU).
Number analyzed (Participants) | 49 | 53
Total number of calls | 123 | 141

2. Primary Outcome: Tobacco Use
Description: Cessation from tobacco use 7-day point prevalent abstinence
Time Frame: 3 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Quitline Treatment As Usual (TAU) | QL Marijuana Check-Up Intervention (QL-MJCU).
Number analyzed (Participants) | 49 | 53
Participants | 14 | 13

3. Primary Outcome: Satisfaction With Treatments
Description: Satisfaction with treatments elicited via outcome survey questions. Question asked, "Overall, how satisfied were you with the Quitline? Would you say…" Answer responses were: VERY SATISFIED; SATISFIED; SOMEWHAT SATISFIED; SOMEWHAT DISSATISFIED; DISSATISFIED; VERY DISSATISFIED; I PREFER NOT TO ANSWER. The outcome measure reported the number of those who responded as being somewhat satisfied or higher.
Time Frame: 3 months
Population: 4 TAU participants did not take any program calls and 1 QJ-MJCU participant withdrew from the study. Their outcomes data were not collected. 15 participants in each group were lost to follow-up and questions were not required to be answered.
Measure: Number; unit: participants
Arm/Group | Standard Quitline Treatment As Usual (TAU) | QL Marijuana Check-Up Intervention (QL-MJCU).
Number analyzed (Participants) | 34 | 37
participants | 28 | 30

4. Primary Outcome: Readiness to Change Marijuana Use
Description: 1-10 scale, where 1 signifies low readiness. On the 3-months post-outcomes survey participants were asked: "On a scale of 1 to 10 where 1 is not at all ready and 10 is very ready, how ready are you to reduce how much cannabis you use?"
Time Frame: 3 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Quitline Treatment As Usual (TAU) | QL Marijuana Check-Up Intervention (QL-MJCU).
Number analyzed (Participants) | 34 | 38
units on a scale | 3.3 (3.4) | 2.9 (2.9)

5. Secondary Outcome: Biochemical Verification of Tobacco Abstinence
Description: Self-administered test of biochemical verification (saliva test) will be sent to participants who self-report tobacco abstinence at 3 month outcomes.
Time Frame: 3 months
Population: Twenty-seven participants reported being quit from tobacco at their follow-up and were mailed a cotinine test kit. Ten of those participants returned results via an emailed photo of their results strip
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Quitline Treatment As Usual (TAU) | QL Marijuana Check-Up Intervention (QL-MJCU).
Number analyzed (Participants) | 3 | 7
Participants | 2 | 5

6. Secondary Outcome: Marijuana Use
Description: Number of days used in the past 30
Time Frame: 3 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Standard Quitline Treatment As Usual (TAU) | QL Marijuana Check-Up Intervention (QL-MJCU).
Number analyzed (Participants) | 34 | 38
days | 23.2 (10.0) | 19.1 (11.8)

ADVERSE EVENTS:
Time Frame: N/A - not assessed
Description: Adverse events were not collected. Upon study initiation, there was a reporting system to collect adverse events; however that was quickly discontinued by the reporting team. The outcomes survey also did not collect information on adverse events; therefore, there is no information regarding adverse events to share.
Arm/Group | Standard Quitline Treatment As Usual (TAU) | QL Marijuana Check-Up Intervention (QL-MJCU).
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-19): https://cdn.clinicaltrials.gov/large-docs/72/NCT04737772/Prot_SAP_000.pdf